CLINICAL TRIAL: NCT02915328
Title: Role of the Type of Carotid Stent and Cerebral Protection on Cerebral Microembolization During Carotid Artery Stenting. A Randomized Study Comparing Carotid Wallstent vs Roadsaver® Stent and Distal vs Proximal Protection.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Principal Investigator, Piero Montorsi, MD, Centro Cardiologico Monzino
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R323/15 - CCM334
Record Dates: First submitted 2016-09-20; First posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Carotid Stenosis
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Stent Roadsaver® +Filterwire EZ™ (Experimental): The arm assess the efficacy of the combination of the stent Roadsaver® with the Filterwire EZ™ protection
  Interventions: Device: Filterwire EZ™; Device: Stent Roadsaver®
- Stent Roadsaver® + MO.MA Ultra (Experimental): The arm assess the efficacy of the combination of the stent Roadsaver® with the MO.MA Ultra protection
  Interventions: Device: MO.MA Ultra; Device: Stent Roadsaver®
- Carotid Wallstent +MO.MA Ultra (Experimental): The arm assess the efficacy of the combination of the Carotid Wallstent with the MO.MA Ultra protection
  Interventions: Device: MO.MA Ultra; Device: Carotid Wallstent
- Carotid Wallstent + Filterwire EZ™ (Experimental): The arm assess the efficacy of the combination of the Carotid Wallstent with the Filterwire EZ™ protection
  Interventions: Device: Filterwire EZ™; Device: Carotid Wallstent

INTERVENTIONS:
Device: Filterwire EZ™
  Arms: Carotid Wallstent + Filterwire EZ™; Stent Roadsaver® +Filterwire EZ™
Device: MO.MA Ultra
  Arms: Carotid Wallstent +MO.MA Ultra; Stent Roadsaver® + MO.MA Ultra
Device: Stent Roadsaver®
  Arms: Stent Roadsaver® + MO.MA Ultra; Stent Roadsaver® +Filterwire EZ™
Device: Carotid Wallstent
  Arms: Carotid Wallstent + Filterwire EZ™; Carotid Wallstent +MO.MA Ultra

SUMMARY:
Stenting is an alternative to traditional surgery in the treatment of carotid stenosis.The intra and/or postprocedural cerebral embolization remains the most frequent complication.

The type of carotid stent and of cerebral protection are the two most important variables potentially affecting the rate of cerebral microembolization. So far there no consensus on the the best stent and cerebral protection.

ELIGIBILITY:
Inclusion Criteria:

significant, unilateral carotid artery stenosis with soft plaque defined as:

* symptomatic patients: > 1.3 m/sec peak systolic velocity and > 50% diameter stenosis by Doppler ultrasound and < 60 hounsfield unit by CT angiography
* asymptomatic patients > 2.5 m/sec peak systolic velocity and > 70% diameter stenosis by Doppler ultrasound and < 60 hounsfield unit by CT angiography

Exclusion Criteria:

* severe cerebral vasculopathy with cognitive impairment
* contraindication to double antiplatelet treatment
* controlateral carotid occlusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
number of microembolization signals (MES) detected with transcranial doppler | intraprocedural
  different phases of carotid stenting (lesion wiring; predilation; stent crossing of the lesion; stent deployment; stent post dilation; device retrieval/deflation

SECONDARY OUTCOMES:
Clinical success | day 2 or day 3 and day 30 complication
  all strokes, major and minor strokes, myocardial infarction
6 month clinical follow up | 6 month
  all strokes, major and minor strokes, myocardial infarction
Doppler ultrasound assesment | day 2 or day 3, 1 month and 6 month
  stent patency and long term restenosis of target carotid artery and target vessel external carotid artery

CONTACTS AND LOCATIONS:
Overall Officials: Piero Montorsi, MD, Principal Investigator — Centro Cardiologico Monzino, IRCCS
Locations (1):
- Centro Cardiologico Monzino, IRCCS, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Montorsi P, Caputi L, Galli S, Ravagnani PM, Teruzzi G, Annoni A, Calligaris G, Fabbiocchi F, Trabattoni D, de Martini S, Grancini L, Pontone G, Andreini D, Troiano S, Restelli D, Bartorelli AL. Carotid Wallstent Versus Roadsaver Stent and Distal Versus Proximal Protection on Cerebral Microembolization During Carotid Artery Stenting. JACC Cardiovasc Interv. 2020 Feb 24;13(4):403-414. doi: 10.1016/j.jcin.2019.09.007. Epub 2020 Jan 29. PMID 32007460